CLINICAL TRIAL: NCT05947656
Title: An Open-label, Non-randomized, Single-arm Pilot Study to Evaluate the Safety and Efficacy of Multiple Pulsed Focused Ultrasound Treatment in Patients With Drug Resistant Temporal Lobe Epilepsy
Brief Title: Evaluation of the NaviFUS System in Drug Resistant Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Genovate-NaviFUS (Australia) Pty Ltd. (Industry)
Collaborators: Genovate Biotechnology Co., Ltd., (Industry); NaviFUS Corporation (Industry)
Responsible Party: Sponsor
Organization: Genovate Biotechnology Co., Ltd., (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNIA22-001
Record Dates: First submitted 2023-06-20; First posted 2023-07-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy, Temporal Lobe; Drug Resistant Epilepsy
Keywords: Focused Ultrasound; Drug Resistant Temporal Lobe Epilepsy; Temporal Lobe Epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: The study consists of two (2) cohorts. Nine (9) eligible patients will be enrolled to each cohort. The only difference between the two cohorts is the overall number of weeks of treatment (2 weeks for Cohort 1 vs. 3 weeks for Cohort 2). The study investigator will advise on which cohort the patients are enrolling into as it will depend on when the patients enter the study. The safety monitoring committee (SMC) will review all safety data for Cohort 1 and confirm that it is safe to proceed with the study before the study treatment for Cohort 2 can start.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Eligible patients in Cohort 1 will receive two (2) FUS treatments per week for two (2) weeks on Day 1, 4, 8 and 11, followed by three (3) safety follow-up visits on Day 36, 64 and 92.
  Interventions: Device: NaviFUS System
- Cohort 2 (Experimental): Eligible patients in Cohort 2 will receive two (2) FUS treatments per week for three (3) weeks on Day 1, 4, 8, 11, 15 and 18, followed by three (3) safety follow-up visits on Day 43, 71 and 99.
  Interventions: Device: NaviFUS System

INTERVENTIONS:
Device: NaviFUS System — NaviFUS System (Neuronavigation-Guided Focused Ultrasound System) is a new non-invasive device, which uses the neuronavigation principle to guide focused ultrasound (FUS) energy precisely delivering through the skull to selected brain tissues without surgery in real-time. In this clinical study, the NaviFUS System is intended to deliver low intensity FUS to generate neuromodulation effects on a predetermined treatment region (one or both of the hippocampi which are associated with seizure), for the treatment for drug-resistant temporal lobe epilepsy (TLE).

SUMMARY:
Participants with drug-resistant epilepsy (DRE) enrolled in this study will receive focused ultrasound (FUS) treatment with the NaviFUS System, guided by the neuronavigation system to evaluate the safety and efficacy of using NaviFUS System. During the treatment, the FUS will electronically scan and target to the assigned zones on one or both of the hippocampi.

The study consists of a 60-day screening period for baseline observation prior to treatment, a FUS treatment period of 2 weeks for Cohort 1 or 3 weeks for Cohort 2 with 2 FUS treatments per week using the NaviFUS System, and a safety follow-up period of 81 days.

DETAILED DESCRIPTION:
Up to 30% of patients with epilepsy are resistant to current anti-seizure medications, i.e. drug-resistant epilepsy (DRE). Resective surgery of the epileptogenic regions is the most effective option to treat patients with DRE. Unfortunately, up to 60% of DRE patients are not suitable for resective surgery.

Neuromodulation approaches are increasingly being utilized in patients with DRE. The current approved techniques use invasive neuromodulation, which require complex neurosurgery and could cause side effects, such as infection, bleeding, and non-target brain tissue damage.

Focused ultrasound is a novel, noninvasive, therapeutic technology with the potential to improve the quality of life and decrease the cost of care for patients with epilepsy. NaviFUS System (a neuro-navigation guided focused ultrasound system) is one of the FUS technologies that uses low-intensity focused ultrasound (LIFU) phased array system to deliver transcranial burst-mode ultrasound energy to induce neuromodulation effect and block signals in a specific area of the brain that cause symptoms of epilepsy such as seizures. The pilot clinical study has demonstrated that NaviFUS System safely delivered LIFU to the seizure onset zone and modulated the neuronal activity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of drug resistant temporal lobe epilepsy (TLE)
2. Patients must experience at least four (4) observable seizures over the 60-day baseline, each on a separate day.
3. Patients have focal-onset seizures with or without secondary generalization.
4. Patients have had at least 24 hours video-electroencephalography (EEG) monitoring and comprehensive epilepsy evaluation confirming TLE.
5. Seizure medication treatment is anticipated to remain stable during the trial, except for rescue medicines or occasional extra doses of ongoing medicines, as required.
6. Patients should be capable of and willing to completing assessments and neuropsychological testing in English either alone or with the help of the study partner (where appropriate), per local guidelines. A study partner is a carer or family member of the patient.
7. Patients and study partner (if applicable) who in the Investigator's opinion are reliable and able to use the seizure diary to record seizure throughout the study and are willing to comply with study procedures and visits.

Exclusion Criteria:

1. Patients who have primary generalized epilepsy or non-epileptic seizures in the last two (2) years.
2. More than two (2) seizure onset zones (foci) (except bitemporal foci) or unknown likely site of seizure onset, as determined by usual clinical, electroencephalography (EEG) and imaging practice.
3. Patients who have experienced tonic-clonic status epilepticus in the three (3) months leading up to enrollment in the study.
4. Presence of devices including but not limited to cardiac pacemaker, implantable cardioverter-defibrillator (ICD), permanent medication pumps, cochlear implants, responsive neurostimulator (RNS) or deep brain stimulation (DBS). Vagus nerve stimulators (VNS) do not represent an exclusion criterion, but settings should be stable throughout the trial.
5. Patients with clips or other metallic implanted objects in the FUS exposure path, except shunts.
6. Patients with more than thirty percent (30%) of the skull area traversed by the sonication pathway covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp at Screening.
7. Patients who have a medical or surgical history of severe systemic disease(s), such as (but not limited to) coronary artery disease, myocardial infarct, progressive heart failure, uncontrolled hypertension or abnormal ECG, severe pulmonary hypertension (pulmonary artery pressure > 90 mmHg), chronic obstructive pulmonary disease (COPD), adult respiratory distress syndrome, hepatic and renal insufficiency (ALT or AST 3 times above normal range; serum creatinine > 1.3 mg/dL), diabetic patients with poor control of blood sugar (HbA1c > 8.5 %) at Screening.
8. History of intracranial hemorrhage.
9. History of multiple strokes, or a stroke within the six (6) months prior to Screening.
10. Patients with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment at any time.
11. Presence of central nervous system (CNS) disease(s) other than epilepsy including but not limited to infections of the CNS (e.g., syphilis, Lyme disease, borreliosis, viral or bacterial meningitis/encephalitis, human immunodeficiency virus [HIV] encephalopathy), cerebral vascular disease, Parkinson's disease, traumatic brain injury, alcoholic encephalopathy within three (3) years prior to Screening.
12. Patients with concurrent major psychiatric disorder, such as schizophrenia or bipolar disorder, severe depression, active suicidal ideation, active psychosis (excluding time-limited postictal psychosis) or psychiatric hospitalization within one (1) year before Screening.
13. Prior diagnosis of cancer within the past two (2) years and evidence of continued malignancy within the past two (2) years (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ prostate cancer with normal prostate-specific antigens post resection).
14. Patients who are not able or willing to tolerate the required prolonged stationary semi-supine position during treatment.
15. Inability to tolerate MRI procedures or contraindication to MRI (e.g. claustrophobia, too large for MRI scanner), including, but not limited to, presence of pacemakers (with the exception of MRI-safe pacemakers), aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or other areas of the body that would contraindicate an MRI scan.
16. Patients who had major surgery six (6) weeks before study enrollment or who are not fully recovered from a surgical procedure or with planned surgery during study period or within fourteen (14) days thereafter.
17. Patients who have received radiofrequency thermocoagulation (RFTC) within two (2) months of Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, nature and severity of adverse events (AEs), serious adverse events (SAEs) and AE of special interest (seizures, headaches, mental state changes, language and memory changes, lethargy/fatigue, and nausea) | Up to 3 months after the last treatment session
  This outcome will be assessed through the review of medical records and participant self-reporting in seizure diary.
Incidence of treatment discontinuation due to AEs and SAEs | Up to 3 months after the last treatment session
Incidence of clinically significant abnormal findings from physical and neurologic examinations | Up to 3 months after the last treatment session
Incidence of clinically significant abnormal vital sign measurements, and abnormal vital signs reported as AEs and SAEs | Up to 3 months after the last treatment session
Incidence of 12-lead electrocardiogram (ECG) with clinically significant abnormal findings | Up to 3 months after the last treatment
Incidence of Magnetic Resonance Imaging (MRI) with clinically significant abnormal findings | Up to 3 months after the last treatment session
  This outcome will be measured at Baseline Visit and 3 months after the last treatment session.
Clinically significant changes in cognitive functions from baseline assessed by Boston Naming Test-Second Edition (BNT-2) | Up to 3 months after the last treatment session
  BNT-2 is a 60-item/picture test to assess the ability to name common objects, with scores ranging from 0 to 60. Higher scores indicate better naming ability.
Clinically significant changes in cognitive functions from baseline assessed by Auditory Naming Test (ANT) | Baseline Visit and 3 months after the last treatment session
  ANT is a 50-item test requiring participants to name a specific item to a description, with scores ranging from 0 to 50. Higher scores indicate better naming ability.
Clinically significant changes in cognitive functions from baseline assessed by Sentence Repetition Test (SRT) | Baseline Visit and 3 months after the last treatment session
  SRT tests immediate memory for sentences of increasing length (1-26 syllables), with scores ranging from 0 to 22. Higher scores indicate better performance.
Clinically significant changes in cognitive functions from baseline assessed by Controlled Oral Word Association Test (COWAT) | Baseline Visit and 3 months after the last treatment session
  COWAT is an oral fluency test in which the participant is required to make verbal associations to different letters of the alphabet by saying as many words as they can think of beginning with a given letter. Greater number of words produced indicates better performance on the test.
Clinically significant changes in cognitive functions from baseline assessed by Wechsler Memory Scale-4 (WMS-4) | Baseline Visit and 3 months after the last treatment session
  WMS-IV measures the ability to learn and remember information presented verbally and visually, with scores ranging from 60 to 140 (mean = 100; standard deviation = 15). Higher scores indicate better performance.
Clinically significant changes in cognitive functions from baseline assessed by Rey Auditory Verbal Learning Test (RAVLT) | Baseline Visit and 3 months after the last treatment session
  RAVLT is a test using a 15-word list to assess non-verbal learning and memory, with scores ranging from 0 to 15. Higher scores indicate better performance.

OTHER OUTCOMES:
Exploratory outcome 1: Change in seizure frequency after FUS treatment compared to baseline | From Baseline Visit until 3 months after the last treatment session
  This outcome will be assessed through the review of medical records and participant self-reporting in seizure diary.
Exploratory outcome 2: Responder rate (defined as at least 50% seizure reduction) | From Baseline Visit until 3 months after the last treatment session
  This outcome will be assessed through the review of medical records and participant self-reporting in seizure diary.
Exploratory outcome 3: Percentage change in days seizure-free | From Baseline Visit until 3 months after the last treatment session
  This outcome will be assessed through the review of medical records and participant self-reporting in seizure diary.
Exploratory outcome 4: Subjective scoring of seizure intensity | From Baseline Visit until 3 months after the last treatment session
  This outcome will be assessed through the review of medical records and participant self-reporting in seizure diary. The seizure intensity (severity) will be scored on a 7-point scale of 1 (very mild) to 7 (very severe).
Exploratory outcome 5: Change in frequency of interictal epileptiform discharges or electrographic seizures on 24 hour ambulatory electroencephalogram (aEEGs) from baseline | Baseline Visit and 3 months after the last treatment session
  This outcome will be measured at Baseline Visit, and 1, 2, and 3 months after the last treatment session.
Exploratory outcome 6: Change in the 31-item Quality of Life in Epilepsy (QOLIE-31) assessment from baseline | Baseline Visit and 3 months after the last treatment session
  The QOLIE-31 includes 31 questions about epilepsy patient's health and daily activities, yielding a composite score from 0 to 100. Higher scores indicate a better quality of life.
  This outcome will be assessed at Baseline Visit, and 1, 2, and 3 months after the last treatment session.
Exploratory outcome 7: Change in Beck Anxiety Inventory (BAI) assessment from baseline | Baseline Visit and 3 months after the last treatment session
  BAI contains 21 questions, each answer being scored on a scale value of 0 (not at all) to 3 (severely). Higher total scores indicate more severe anxiety symptoms.
  This outcome will be assessed at Baseline Visit, and 1, 2, and 3 months after the last treatment session.
Exploratory outcome 8: Change in Beck Depression Inventory-2 (BDI-2) assessment from baseline | Baseline Visit and 3 months after the last treatment session
  BDI-2 consists of 21 questions, and a value of 0 to 3 is assigned for each answer, ranging in intensity. Higher total scores indicate more severe depressive symptoms.
  This outcome will be assessed at Baseline Visit, and 1, 2, and 3 months after the last treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence O'Brien, Prof., Principal Investigator — The Alfred
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No